CLINICAL TRIAL: NCT05049005
Title: Dietary Approaches for Improving Engagement, Diet Quality, and Weight Loss in Young Adults
Brief Title: Alternative Dietary Approaches Online to Promote Tracking
Acronym: ADOPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-0491
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-03

CONDITIONS: Diet Quality; Weight Loss
Keywords: Adherence, diet tracking, diet goals
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RED FOOD Intervention Group (Active Comparator): Participants in the RED FOOD group will be taught a simplified way of identifying high-calorie foods (red foods) and reducing them using the Traffic Light Diet. Limiting the number of red foods consumed is a simple way to reduce calories without having to track calories. Participants in this group will use the study website to track their red foods and will be given a daily red food limit base on their baseline weight and will track their red foods on the study website daily. Participants will be recommended to enter their red foods at least once per day (at which time they would enter all red foods for the day), but ideally multiple times per day to reduce errors associated with recall.
  Interventions: Behavioral: Simplified dietary tracking
- GREEN FOOD Intervention Group (Experimental): Participants in the GREEN FOOD group will be taught a simplified way of identifying low-calorie foods (green foods) and maximizing them using the Traffic Light Diet. Maximizing the number of green foods consumed is a simple way to reduce dietary energy density while allowing for consumption of a satisfying amount (i.e. weight and volume) of food. Maximizing green food consumption may simultaneously reduce red food consumption, thereby reducing calorie intake and promoting greater diet quality than red food reduction alone. Participants in this group will also use the study website to track their green foods and will be given a daily green food goal based on their baseline weight and will track their green foods on the study website daily. Participants will be recommended to enter their green foods at least once per day (at which time they would enter all green foods for the day), but ideally multiple times per day to reduce errors associated with recall.
  Interventions: Behavioral: Simplified dietary tracking

INTERVENTIONS:
Behavioral: Simplified dietary tracking — Mobile-delivered nutrition program using simplified dietary monitoring with a focus on weight loss.

SUMMARY:
Purpose: Compare the efficacy of two 3-month Internet-based interventions that use a simplified strategy for monitoring of dietary intake among young adult men and women with overweight or obesity.

Participants: Young adult men and women who are between the ages of 18-35 years (N=75) and who currently have overweight or obesity (BMI between 25 and 50 kg/m^2).

Procedures (methods): This is a randomized controlled trial comparing the efficacy of two Internet-based dietary interventions among 75 young adult men and women who currently have overweight or obesity. Both interventions will use simplified monitoring of dietary intake using an approach based on the Traffic Light Diet. One intervention will target a reduction in intake of red foods (high-calorie, high-fat foods) and tracking of red foods in the study website. The other intervention will target an increase in intake of green foods (low-calorie, healthy foods) and tracking of green foods in the study website. Components of both interventions include (1) personalized goals for red/green food intake, (2) weekly tailored feedback, and (3) weekly lessons delivered via smartphone.

DETAILED DESCRIPTION:
The primary objective of the study is to test two approaches for dietary self-monitoring among young adults with overweight/obesity. Thus, all participants will receive an Internet-based dietary intervention that includes evidence-based lessons focused on dietary change, behavioral skills training, and frequent weighing. The only difference between the two groups will be the types of foods participants are instructed to self-monitor and the dietary goals participants are given. Young adult men and women (N=75) will be randomly assigned, with equal probability, to one of two groups:

1. Red food reduction intervention (RED FOOD): An Internet-based dietary intervention delivered via REDCap; weekly self-report of weight and daily red food monitoring using a mobile-optimized study website.
2. Green food promotion intervention (GREEN FOOD): An Internet-based dietary intervention delivered via REDCap; weekly self-report of weight and daily green food monitoring using a mobile-optimized study website.

During the 3-month Internet-based dietary intervention, participants will receive an email at the beginning of each week with a link to a REDCap page that will ask them to self-report their weight. They will then be directed via REDCap to their tailored feedback summaries based on their self-reported weight data and the dietary monitoring data that is pulled from the study website. After reading their feedback, participants will be directed to a weekly lesson in REDCap. Participants will be encouraged to login to the study website every day to self-monitor red or green foods, depending on their intervention group. Participants will receive a unique username and password to login to the study website. Each intervention component is described in more detail below.

Intervention Components:

Participant goals: Participants will be assigned a dietary goal based on their baseline weight. Participants will be able to view their daily dietary goal (number of red foods per day in RED FOOD and number of green foods per day in GREEN FOOD) on the study website. Participants' dietary goals will be based on their intervention group. Participants will not receive specific goals for weighing or physical activity. However, all participants will be recommended to weigh frequently throughout the week, as research has shown this is best for successful weight loss. Participants will self-report their weight online via REDCap once per week.

Weekly feedback: Participants will receive tailored feedback summaries via REDCap weekly. Participants will receive an email to self-report their weight in REDCap, after which they will be directed to their feedback page. The feedback message will include feedback based on participants' number of days tracking diet, progress toward their dietary goal, and self-reported weight for the week.

Lessons: Lessons will be updated weekly and made available in REDCap. Lesson content will focus on specific areas of diet or eating behavior which participants could focus on changing over the next week. Behavioral topics typically included in behavioral weight control programs will be incorporated into the lessons including problem solving, planning ahead, and stimulus control. Participants will be directed to the REDCap lesson after reviewing their weekly feedback message.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 25 and 50 kg/m^2
* English-speaking and writing
* Own a smartphone with an active data and text messaging plan
* Own a bathroom scale or willing to purchase a bathroom scale prior to the study start date
* Willing to be randomized to either group

Exclusion Criteria:

* Type I or Type 2 diabetes
* Currently participating in another nutrition or weight loss program
* Lost 10 or more pounds (and kept it off) in the last 6 months
* Currently taking weight loss medications
* Currently pregnant, pregnant within the past 6 months, or planning to become pregnant in the next 6 months
* Serious current physical disease (i.e. heart disease, stroke, cancer, or renal disease) for which physician supervision of diet and exercise prescription is needed
* Physical problems that limit the ability to exercise daily
* History of clinically diagnosed eating disorder
* Report a past diagnosis of or current symptoms of alcohol or substance dependence
* Diagnosis of schizophrenia or bipolar disorder
* Hospitalization for a psychiatric diagnosis within the last year
* Currently living with another study participant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Adherence to dietary tracking | 3 months
  Adherence will be assessed via frequency of dietary monitoring. Each food entry will be time-stamped and automatically captured by the study website interface. Frequency of dietary monitoring will be defined as the total number of days during the 3-month intervention that participants tracked breakfast or lunch AND dinner, which will be considered a full (versus partial) day of tracking.
Adherence to dietary goals | 3 months
  Adherence will be measured as the total number of full days of tracking (i.e. breakfast or lunch AND dinner) during which participants met their dietary goal. Non-adherence will be assumed for partial days of tracking, or days where participants did not track.

SECONDARY OUTCOMES:
Percent weight loss | 3 months
  Percent weight loss (PWL) from baseline to 3 months will be calculated using the following formula, which results in increasingly negative values as weight declines: ((weight at 3 months - baseline weight)/baseline weight)*100
Change in Dietary intake | Baseline, Month 3
  Assessed using using the Automated Self-Administered 24-Hour Recall (ASA24). This online system guides participants through a multi-pass recall of foods eaten over the previous 24 hours. Intake will be measured twice (one weekday and one weekend day) at each time point to provide the most accurate representation of typical consumption. The system creates researcher reports of intake that include total energy intake, macronutrients, and micronutrients.
Change in Diet quality | Baseline, Month 3
  The Healthy Eating Index (HEI)-2015 will be used to assess diet quality based on the major dietary recommendations of the 2015 Dietary Guidelines for Americans (DGA). The HEI-2015 consists of 13 component scores, including: total fruit, whole fruit, total protein foods, total vegetables, greens and beans, whole grains, dairy, seafood and plant proteins, fatty acids, sodium, refined grains, added sugars, and saturated fats. The summation of the 13 component scores ranges from 0 to 100, with higher scores indicating closer compliance with the 2015 DGA.

OTHER OUTCOMES:
Change in Restraint, Disinhibition, Hunger | Baseline, Month 3
  Assessed with the 51-item Three-Factor Eating Questionnaire. The cognitive restraint scale (21 items) measures conscious attempts to monitor and regulate food intake, the disinhibition scale (16 items) measures uncontrolled eating in response to cognitive or emotional cues, and the perceived hunger scale (14 items) measures the extent to which respondents experience feelings of hunger in their daily lives. Higher scores indicate higher levels of cognitive restraint, disinhibition, and perceived hunger. Each item scores either 0 or 1 point, therefore, minimum scale scores are 0-0-0 while maximum scale scores are 21-16-14.
Change in Self-Regulation (eating behaviors) | Baseline, Month 3
  Assessed using the 26-item Eating Behavior Inventory (EBI). The EBI is a self-report instrument for assessing behaviors that have been associated with weight loss, e.g., self-monitoring of food intake and of weight, refusing offers of food, eating at only one place, shopping from a list, eating in response to emotions. Each item is rated with a 5-point Likert scale ranging from 1 (Never or hardly ever) to 5 (Always or almost always). Items are scored (after reverse-coding certain items) such that higher scores always reflect eating patterns that are more favorable for weight control. Scores range from 26-130.
Change in Self-Regulation (global) | Baseline, Month 3
  Assessed using the 31-item Short Self-Regulation Questionnaire (SSRQ). The SSRQ is a self-report measure of the ability to regulate behavior to achieve one's goals. The SSRQ consists of one scale and participants respond using a 5-point Likert scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree). Items are scored (after reverse-coding certain items) such that higher scores reflect greater self-regulation capacity. Scores range from 31-155.
Change in Self-Efficacy (diet) | Baseline, Month 3
  Assessed using the 20-item Weight Efficacy Lifestyle (WEL) Questionnaire. The WEL consists of five scales: negative emotions, availability, social pressure, physical discomfort, and positive activities. Scales are measured using ten response options ranging from 0 (not confident) to 9 (very confident). Higher scores indicate greater confidence in one's ability to control weight by resisting overeating in certain tempting situations. Subscale scores range from 0 to 36, and total score ranges from 0 to 180.

CONTACTS AND LOCATIONS:
Overall Officials: Julianne M Power, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Weight Research Program, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No